CLINICAL TRIAL: NCT00200798
Title: Pharmacokinetics and Drug Interactions With Milk Thistle
Brief Title: An Assessment of Milk Thistle Pharmacokinetics and Drug Interactions
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: John S. Markowitz, Pharm.D., MUSC
Other Study IDs: R21AT002817-01 (NIH); R21AT002817-01 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: Milk Thistle; Silymarin; pharmacokinetics; drug interactions; Normal volunteers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma & urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is accumulating evidence from various sources that extracts from the milk thistle plant can be useful in the treatment of a variety of liver ailments as well as other disorders. This investigation will essentially be composed of two individual normal volunteer studies of milk thistle. The first study will assess the rate and extent of absorption of components of a standardized botanical extract obtained from the milk thistle plant. This first study is termed a bioavailability study. This investigation will take approximately 8 weeks and involve 10 clinic visits. Secondly, a drug interaction study will be performed. This is an assessment study of the potential for this botanical extract to interact with other prescription or over-the-counter medications. This study is also expected to take approximately 8 weeks but will involve 18 clinic visits. In both studies all subjects will receive the same milk thistle supplement and no placebo will be administered.

DETAILED DESCRIPTION:
BIOAVAILABILTY STUDY:

1. Clinical Protocol

Screening/Informed Consent: Sixteen subjects will be recruited for the clinical protocol. All protocols, consent forms, and HIPAA forms shall be IRB-approved prior to initiating any study procedure or recruitment. At a screening/informed consent visit, the study design, purposes and inclusion/exclusion criteria will be explained to each prospective subject. Written informed consent will be obtained prior to commencing any study procedures. After informed consent is obtained, medical examinations will be performed along with baseline serum chemistries, complete blood count, electrocardiogram, urinalysis, urine drug screen, nicotine/cotinine, and urine pregnancy test (females). Subjects will be asked about their diets including alcohol use and the use of herbal medications/dietary supplements. If a potential subject has been consuming any herbal or dietary supplements a two-week period of abstinence from supplement use will be necessary before beginning the study. Additionally, subjects will refrain from use of honey or propolis-containing products (due to presence of chrysin and potential assay interference), and artichokes, or artichoke-containing foods that also contain taxifolin (a constituent found in MT).

Single- and Multiple-Dose Silymarin Pharmacokinetics: Subjects will arrive at the MUSC GCRC in the morning where they will remain for approximately 10-hours for each of 4 separate blood drawing phases of the study. After checking in, and under medical supervision, a modification of a modified Treatment Emergent Symptoms Scale (TESS) will be administered and a registered nurse will place an indwelling venous catheter in each subject's arm to facilitate serial blood sampling. At 8 AM after urinary void and collection of an aliquot for creatinine analysis, subjects will take one 175 mg capsule of MT standardized to 80% SM (140 mg of SM). The rationale for product choice is discussed below. Subjects will be in a fasted state for 4 hours following MT administration to reduce any effect of food on absorption. A total of 12 blood samples (10 ml each) will be taken over the next 24-hour period. All samples will be drawn in heparinized tubes and stored on ice until centrifugation at 4°C. As flavonoids are notorious for their instability in biological matrices, no sample will remain on ice for longer than 15 minutes prior to centrifugation. Time points of blood collection will be immediately prior to the dose of MT (0 time point), and at 0.5 hours, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12, and 24 hours. A second TESS will be administered to the subjects 2 hours post-dosing, at a time generally expected to represent silybin Cmax. Subjects will be asked to return for 4 brief visits for collection of single blood samples through a separate venipuncture at time points of 24, 36, and 48 hours. This extended sampling will provide adequate PK data to determine Cmax, AUC, terminal t1/2, and Clo of SM flavonoids. Standard meals will be served by the registered dietician at the GCRC and will not include any other sources of flavonoids. The composition and amount of food eaten throughout the day will be recorded. Plasma will be acidified with 10 ml of 1M acetic acid/ml plasma and frozen immediately at -70°C. This single dose assessment of silymarin pharmacokinetics will be conducted at three dosage levels of MT supplement in an attempt to span the usual therapeutic range of MT and will be performed on three distinct occasions separated by no less than a 7-day wash-out period. The doses of MT used will be 175 mg, 350 mg and 525 mg administered orally with 200 mL of water as one, two, and three capsules, respectively. Again, these doses as well as product could be changed if a more standardized supplement is made available through NIH/NCCAM or some other source. The highest dose of MT supplement proposed for oral administration, 525 mg (420 mg SM) does not pose any undue risk to subjects since SM doses of 420 mg to 800 mg has been administered to many patients with hepatic dysfunction in clinical trials with few side effects reported (NLM, 2000; Saller et al., 2001).

Following the last single dose assessment and an ensuing 7-day minimum wash-out period, subjects will initiate treatment of a 28-day treatment exposure to the MT supplement 175 mg (140 mg SM) at the generally recommended and clinically studied dosage of one capsule thrice daily (NLM, 2000). A 28-day course is selected to assure steady-state is reached and to surpass the duration of any other published pharmacokinetic studies of SM in human subjects which have generally been of brief duration. In addition, this extended dosing assessment will allow for the gathering of pilot data on the antioxidant potential of SM via measurements of urinary isoprostanes. Finally, an assessment of treatment-emergent adverse effects and tolerability will be made. Subjects will report to the outpatient GCRC on 4 separate occasions to pick up a 7-day supply of SM at which time a TESS will be administered. At the initial visit to the GCRC to obtain the first week's supply of MT, subjects will provide a urine sample for baseline measurement of urinary isoprostanes and creatinine. After 28 days of treatment subjects will report to the GCRC for the determination of steady-state concentrations of SMs in plasma and urine. A blood draw will be performed immediately prior to dosing with the MT (Ctrough) and 0.5, 1.0, 2.0, 3.0 and 4.0 and 8.0 following MT dosing. Based upon available published data, these timepoints should be sufficient to capture the (Cmax) for all flavonoids of interest despite interindividual variability. Additionally, subjects will provide a morning urine sample for analysis of urinary isoprostane and creatinine.

Follow-Up: Subjects will return 7 days following the final blood draw to have a follow-up serum chemistry and complete blood count (CBC) performed to provide an additional assurance of subject safety. We will also perform a final assessment of adverse events using the TESS scale.

DRUG INTERACTION ASSESSMENT:

1. Clinical Protocol for Drug Interaction Assessment

An outline of the proposed clinical study to determine the drug interaction potential of silymarin

Assessing Cytochrome P450 Activity in vivo with Probe Drugs

Probe substrate compounds for the major CYP enzymes are available to assess genetic, environmental, and ethnic differences in enzyme activity. In the last 2 years our research group has published 7 full research reports utilizing probe drug methodology in assessing botanical-drug interactions. These studies were likewise funded by NCCAM, had an excellent safety record, and were performed within the MUSC GCRC.

Probe compounds can be initially administered to subjects in the absence of suspected enzyme inhibitors or inducers and the parent drug or drug: metabolite ratios measured in plasma and urine to reflect enzyme activity. This assessment can then be repeated in the presence of a suspected inhibitor or inducer and comparisons can be made. In this manner, specific enzyme inhibitory or inductive effects can be elucidated, documented, and generalized to other similar substrates. In this study, by using the selected probe substrates alprazolam (CYP3A4), dextromethorphan (CYP2D6), tolbutamide ([TOL] CYP2C9) and caffeine (CYP1A2), we will assess the ability of MT/SM to selectively alter one or more of the major drug metabolizing enzymes responsible for the metabolism of > 80% of all therapeutically used drugs.

We propose to use these validated and widely accepted methods to evaluate the drug-interaction potential of a characterized MT supplement. A clinical protocol, using 16 normal volunteers, will evaluate the potential to inhibit or induce CYP3A4, CYP1A2, CYP2C9, and the potential to inhibit CYP2D6 (a non-inducible isoform). Test doses of these four safe probe drugs will be administered at baseline (before treatment with MT) and after a 14-day treatment period. Changes in the pharmacokinetics of these probe drugs will indicate the degree of specific enzyme inhibition or induction, respectively. These data will be used to evaluate the effects of combining a standardized MT supplement with other drugs that are substrates for the CYP enzymes studied.

Screening/Informed Consent: Sixteen subjects will be recruited for the clinical protocol and replacements will be recruited if necessary for 16 subjects to complete the protocol. Screening and a separate informed consent process will take place as in the pharmacokinetic study previously described with the following exceptions: Subjects will be genotyped to determine if they are poor metabolizers of CYP2D6 substrates. Subjects will also be asked about adverse events according to a Treatment Emergent Symptoms Scale ([TESS] Zhang et al., 2001) to determine if any symptoms are present prior to administration of the MT supplement. Subjects will be asked about their diets including alcohol use and the use of herbal medications/dietary supplements. If a potential subject has been consuming any herbal or dietary supplements a two week period of abstinence from supplement use will be necessary before beginning the next study phase.

Baseline CYP profile: Subjects will return to the GCRC at a specified time in the morning prior to probe drug administration. In the morning, an indwelling venous catheter will be placed in each subject's arm to facilitate serial blood sampling. At 8AM, after urinary void, subjects will be asked to take simultaneous single oral doses of 2 mg ALPZ, 100 mg CAF, 100 mg TOL, and 30 mg DM. At this time, a urine collection will commence for the first eight hours of the visit. A total of 11 blood samples (10 ml each) will be taken over a 12-hour period. Time points of blood collection will be immediately before drug administration, and at 0.5 hours, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, and 12 hours. Additionally, the subjects will be asked to return for 4 more brief visits for collection of single blood samples through a separate venipuncture at time points of 24, 36, and 48 hours. This extended sampling will provide adequate pharmacokinetic data to determine Cmax, AUC, terminal t1/2, and Clo of all probe drugs. To reduce any potential variability in drug absorption due to food, the subjects will be in a fasted state for 4 hours following probe drug administration. Standard meals will be served by the registered dietician at the GCRC and will not include grapefruit, artichoke products, or CAF. The composition and amount of food eaten throughout the day will be recorded.

MT Treatment Period: Subjects will commence treatment with the MT supplement 175 mg (140 mg SM) one capsule three times daily (8AM, 12 noon, 8PM) for a period of 14 days. Subjects will be supplied with pre-loaded medication organizers containing the daily doses of MT to promote compliance with the regimen. Subjects will be asked to return to the study site for 4 pre-scheduled appointments during this time for capsule counts, to discuss compliance with dietary restrictions, and for monitoring of adverse events.

Post-MT CYP profile: Subjects will return to the GCRC for this phase of the study. Subjects will check in the morning prior to a repeat dosing of probe medications. The profiling of CYP3A4, CYP2D6 and CYP1A2 will be performed exactly as described for the baseline phase with the exception that for the first 24 hours subjects will continue their previous schedules of dosing with the MT supplement. The doses of probe drugs will coincide with the 8AM dose of MT so that they will be taken concomitantly. Blood and urine sampling times will be identical. As in the baseline phase, subjects will be in a fasted state for 4 hours following probe drug administration. Additionally, subjects will be served identical meals at the same timepoints as in the baseline phase.

Follow-Up: Subjects will return 7 days following the final blood draw to have a follow-up serum chemistry and complete blood count (CBC) performed to provide an additional assurance of subject safety. We will also perform a final assessment of adverse events using the TESS scale.

Probe Drugs: Alprazolam (ALPZ), dextromethorphan (DM), tolbutamide (TOL) and caffeine (CAF)

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-45 years old
* Race or ethnicity: no restrictions
* Health status: subjects must have no clinically significant diseases or clinically significant abnormal laboratory values as assessed during the screening medical history, physical exam, and laboratory evaluations.
* Must have no history of significant psychiatric illness or substance use.
* Written Informed Consent as well as Health Insurance Portability and Accountability Act (HIPAA) authorization forms must be signed by the eligible subject prior to the initiation of any study procedures.

Exclusion Criteria:

Any of the following conditions are cause for exclusion and/or discontinuation from the study:

* The presence of any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion.
* A positive urine pregnancy test
* The use of oral contraceptives
* The lack of use of acceptable barrier methods of birth control unless abstinent
* The use of any concomitant medication including herbal medications, over-the-counter (OTC) supplements, or a history of hypersensitivity to DM, ALPZ, TOL, or caffeine (CAF) and any history of sensitivity to milk thistle or any of its components.
* Subjects genotyped as poor metabolizers of CYP2D6 at screening
* Active smoking or use of CAF containing beverage (coffee, certain colas) for one week prior and during the study period due to known effects on CYP1A2 activity.
* Subjects expressing inability to conform to dietary restrictions required for the study
* The use of any illicit drugs or habitual consumption of large quantities of ethanol (> 3 drinks/day)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S. Markowitz, Pharm.D., Principal Investigator — Medical University of South Carolina; Thomas W Uhde, MD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, GCRC, Charleston, South Carolina, United States